CLINICAL TRIAL: NCT01333397
Title: A Phase II, Double Blind, Randomised, Placebo and Active Comparator Controlled Study to Assess the Safety and Efficacy of Three Doses of Dysport RU (20 U, 50 U, and 75 U) Administered as a Single Treatment Cycle to Improve the Appearance of Moderate to Severe Glabellar Lines
Brief Title: Safety and Efficacy Study of Dysport RU and Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y-52-52120-146; 2010-019085-82 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dysport RU 20 U (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Dysport RU 50 U (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Dysport RU 75 U (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Dysport (Azzalure) 50 U (Active Comparator)
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — I.M. (in the muscle) injection on day 1 (single treatment cycle)
  Other Names: AbobotulinumtoxinA (DysportRU®)
  Arms: Dysport RU 20 U; Dysport RU 50 U; Dysport RU 75 U
Biological: Botulinum toxin type A — I.M. on day 1 (single treatment cycle)
  Other Names: AbobotulinumtoxinA (Azzalure®)
  Arms: Dysport (Azzalure) 50 U
Drug: Placebo — I.M. on day 1 (single treatment cycle)
  Arms: Placebo

SUMMARY:
The primary objective is to assess the dose response versus placebo of a single treatment of Dysport RU (Dysport RU, Ready to Use, for injection), for the improvement in appearance of moderate to severe glabellar lines at maximum frown.

ELIGIBILITY:
Inclusion Criteria:

* Female between 30 - 60 years of age
* Moderate to severe vertical glabellar lines at maximum frown at baseline

Exclusion Criteria:

* Silicone injections into the upper face
* Any prior treatment with fillers (e.g. collagen-type implants) skin abrasions or photorejuvenation within the previous 12 months
* Any planned facial cosmetic surgery during the study period
* A history of ablative skin resurfacing of the area to be treated during the study.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (8):
- France (4):
  - Private practice, Bordeaux
  - Private practice, Cannes
  - Private practice, Juan-les-Pins
  - Private practice, Paris
- Germany (4):
  - Charité hospital, Berlin
  - Private clinic, Dresden
  - Private clinic, Munich
  - Private clinic, Starnberg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was performed as a multicentre study at eight investigational sites in France and Germany. Date of first enrolment: 30-Mar-2011 and Date of last completed: 27-Sep-2011.
Pre-assignment Details: A total of 178 patients were screened. 2 patient did not meet the entry criteria. 176 patients were randomized.Patients were randomized into 5 groups.
Groups:
- Placebo: Intramuscular injections on Day 1 (total injection volume of 0.25 ml divided into five intramuscular injections of 0.05 mL per injection each of which was injected into five pre-defined sites across the glabellar region) (single treatment cycle)
- Dysport NG 20 U: Botulinum type A toxin (Dysport RU), Intramuscular injections on Day 1 in the muscle (total injection volume of 0.25 ml divided into five intramuscular injections of 0.05 mL per injection each of which was injected into five pre-defined sites across the glabellar region) (single treatment cycle)
  Ready to Use (RU)
- Dysport NG 50 U; Dysport NG 75 U: Botulinum type A toxin (Dysport RU), Intramuscular injections on Day 1 in the muscle (total injection volume of 0.25 ml divided into five intramuscular injections of 0.05 mL per injection each of which was injected into five pre-defined sites across the glabellar region) (single treatment cycle)
- Dysport 50 U: Botulinum type A toxin (Azzalure), Intramuscular injections on Day 1 (total injection volume of 0.25 ml divided into five intramuscular injections of 0.05 mL per injection each of which was injected into five pre-defined sites across the glabellar region) (single treatment cycle)
Period: Overall Study
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Started | 35 | 36 | 35 | 35 | 35
Completed | 34 | 36 | 35 | 34 | 35
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dysport NG 20 U; Dysport NG 50 U; Dysport NG 75 U: Botulinum type A toxin (Dysport RU), Intramuscular injections on Day 1 in the muscle (total injection volume of 0.25 ml divided into five intramuscular injections of 0.05 mL per injection each of which was injected into five pre-defined sites across the glabellar region) (single treatment cycle)
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U | Total
Number analyzed (Participants) | 35 | 36 | 35 | 35 | 35 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (6.4) | 46.7 (8.4) | 48.1 (6.9) | 47.9 (6.0) | 47.0 (6.6) | 47.3 (6.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 35 | 36 | 35 | 35 | 35 | 176
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 2 | 0 | 2 | 1 | 5
  Not Hispanic or Latino | 35 | 34 | 35 | 33 | 34 | 171
Race/Ethnicity, Customized [Number; unit: participants]
  White | 35 | 36 | 35 | 35 | 35 | 176

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects as Responders in the ILA (Using Validated 4-point Photographic Scale) and the SSA of Glabellar Lines at Maximum Frown
Description: Investigator's live assessment (ILA), subject's self assessment (SSA), Next Generation (NG)
  4-point photographic scale: Investigator's live assessment: None - 0; Mild - 1; Moderate - 2; Severe - 3;
  4-point photographic scale: Subject's Self assessment: No wrinkles - 0; Mild wrinkles - 1; Moderate wrinkles - 2; Severe wrinkles - 3;
  A responder at maximum frown was defined as a subject having a severity grade of none or mild at maximum frown on Day 29 and a severity grade of moderate or severe at maximum frown at Visit 2.
Time Frame: Day 29
Population: Intent-to-Treat Population: The intent-to-treat (ITT) population included all randomised subjects who received study treatment, regardless of the actual amount injected. N'=number of subjects with assessment
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U
Number analyzed (Participants) | 34 | 36 | 35 | 33
percentage of subjects
  ILA (N'=34,36,35,33) | 0 | 88.9 | 91.4 | 87.9
  SSA (N'=34,36,35,33) | 2.9 | 91.7 | 85.7 | 81.8
Statistical Analysis 1: Comparison: Placebo vs Dysport NG 20 U; ILA - Dysport NG 20 U Vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Dysport NG 50 U; ILA - Dysport NG 50 U Vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Dysport NG 75 U; ILA - Dysport NG 75 U Vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Placebo vs Dysport NG 20 U; SSA - Dysport NG 20 U Vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 5: Comparison: Placebo vs Dysport NG 50 U; SSA - Dysport NG 50 U Vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 6: Comparison: Placebo vs Dysport NG 75 U; SSA - Dysport NG 75 U Vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Percentage of Subjects as Assessed as Responders, by Both Investigator's Live Assessment and the Subject's Self-assessment at Maximum Frown.
Description: A responder at maximum frown was defined as a subject having a severity grade of none or mild at maximum frown on the visit day and a severity grade of moderate or severe at maximum frown at Visit 2.
Time Frame: Day 29
Population: ITT Population; Day 29 (N'=34,36,35,33,35); N'= number of subjects with an Investigator's live assessment and a subject's self assessment of glabellar lines at maximum frown for the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 34 | 36 | 35 | 33 | 35
percentage of subjects | 0 | 86.1 | 85.7 | 81.8 | 77.1

3. Secondary Outcome: Percentage of Subjects as Responders at Maximum Frown as Measured by the Investigator's Live Assessment.
Time Frame: Days 8, 15, 57, 85 and 113
Population: ITT Population; N'=number of subjects with an Investigator's live assessment of glabellar lines at maximum frown for the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U
Number analyzed (Participants) | 34 | 36 | 35 | 35
percentage of subjects
  ILA: Day 8 (N'=34,36,35,35) | 0 | 77.8 | 80.0 | 82.9
  ILA: Day 15 (N'=33,36,35,35) | 3.0 | 80.6 | 94.3 | 91.4
  ILA: Day 57 (N'=33,35,34,34) | 0 | 77.1 | 79.4 | 82.4
  ILA: Day 85 (N'=34,33,34,32) | 0 | 48.5 | 58.8 | 75.0
  ILA: Day 113 (N'=34,36,35,34) | 0 | 22.2 | 42.9 | 55.9

4. Secondary Outcome: Percentage of Subjects as Responders at Maximum Frown as Measured by the Subject's Self-assessment.
Time Frame: Days 8, 15, 57, 85 and 113
Population: ITT Population; N'= number of subjects with a subject's self assessment of glabellar lines at maximum frown for the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U
Number analyzed (Participants) | 34 | 36 | 35 | 35
percentage of subjects
  SSA: Day 8 (N'=34,36,35,35) | 2.9 | 66.7 | 65.7 | 74.3
  SSA: Day 15 (N'=33,36,35,35) | 3.0 | 80.6 | 82.9 | 80.0
  SSA: Day 57 (N'=34,35,34,34) | 0 | 80.0 | 67.6 | 82.4
  SSA: Day 85 (N'=34,35,34,32) | 0 | 57.1 | 47.1 | 62.5
  SSA: Day 113 (N'=34,36,35,34) | 0 | 36.1 | 34.3 | 52.9

5. Secondary Outcome: Percentage of Subjects Assessed as Responders, by Both the Investigator's Live Assessment and the Subject's Self-assessment at Maximum Frown.
Time Frame: Days 8, 15, 57, 85 and 113
Population: ITT Population; N'= number of subjects with an Investigator's live assessment and a subject's self assessment of glabellar lines at maximum frown for the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 34 | 36 | 35 | 35 | 35
percentage of subjects
  Day 8 (N'=34,36,35,35,35) | 0 | 61.1 | 62.9 | 74.3 | 51.4
  Day 15 (N'=34,36,35,35,34) | 0 | 75.0 | 82.9 | 80.0 | 67.6
  Day 57 (N'=34,35,34,34,34) | 0 | 74.3 | 67.6 | 79.4 | 64.7
  Day 85 (N'=34,33,34,32,34) | 0 | 42.4 | 44.1 | 62.5 | 38.2
  Day 113 (N'=34,36,35,34,35) | 0 | 19.4 | 34.3 | 41.2 | 25.7

6. Secondary Outcome: Percentage of Subjects as Responders at Rest as Measured by the Investigator's Live Assessment.
Description: A responder at rest was defined as a subject having a severity grade of none or mild at rest on the visit day and a severity grade of moderate or severe at rest at Visit 2.
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: ITT Population; N'= number of subjects with an Investigator's live assessment of glabellar lines at rest of moderate or severe at Baseline and with an assessment at the given post-Baseline visit;
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U
Number analyzed (Participants) | 18 | 17 | 13 | 14
percentage of subjects
  ILA: Day 8 (N'=18,17,13,14) | 11.1 | 70.6 | 76.9 | 71.4
  ILA: Day 15 (N'=18,17,13,14) | 11.1 | 70.6 | 92.3 | 78.6
  ILA: Day 29 (N'=18,17,13,14) | 5.6 | 82.4 | 76.9 | 85.7
  ILA: Day 57 (N'=17,16,13,14) | 11.8 | 81.3 | 76.9 | 78.6
  ILA: Day 85 (N'=18,17,12,14) | 5.6 | 82.4 | 75.0 | 64.3
  ILA: Day 113 (N'=18,17,13,14) | 11.1 | 52.9 | 53.8 | 57.1

7. Secondary Outcome: Percentage of Subjects as Responders at Maximum Frown on Day 29 Who Remain Responders
Description: as for outcome 2
Time Frame: Day 113
Population: ITT Population; N'=number of responders at Day 29
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 1 | 33 | 32 | 29 | 29
percentage of subjects
  ILA: Day 29 (N'=0,32,32,29,27) | 0 | 25.0 | 46.9 | 65.5 | 40.7
  SSA: Day 29 (N'=1,33,30,27,29) | 0 | 36.4 | 40.0 | 63.0 | 34.5

8. Secondary Outcome: Percentage of Subjects With a Reduction of Two or More Grades in the Severity of Glabellar Lines at Maximum Frown as Measured by the Investigator's Live Assessment
Description: A reduction of two or more grades in the severity of glabellar lines at maximum frown was a change from Visit 2 severity of glabellar lines from severe to mild/none or from Visit 2 severity of moderate to none after treatment as measured by the Investigator's live assessment
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: ITT Population; N'= number of subjects with an Investigator's live assessment of glabellar lines at maximum frown for the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 34 | 36 | 35 | 35 | 35
percentage of subjects
  ILA: Day 8 (N'=34,36,35,35,35) | 0 | 30.6 | 45.7 | 45.7 | 31.4
  ILA: Day 15 (N'=33,36,35,35,34) | 0 | 50.0 | 62.9 | 57.1 | 50.0
  ILA: Day 29 (N'=34,36,35,33,35) | 0 | 55.6 | 68.6 | 63.6 | 57.1
  ILA: Day 57 (N'=33,35,34,34,34) | 0 | 34.3 | 47.1 | 44.1 | 41.2
  ILA: Day 85 (N'=34,33,34,32,34) | 0 | 24.2 | 29.4 | 31.3 | 26.5
  ILA: Day 113 (N'=34,36,35,34,35) | 0 | 13.9 | 14.3 | 20.6 | 8.6

9. Secondary Outcome: Percentage of Subjects With a Reduction of Two or More Grades in the Severity of Glabellar Lines at Rest as Measured by the Investigator's Live Assessment
Description: A reduction of two or more grades in the severity of glabellar lines at rest was a change from Visit 2 severity of glabellar lines from severe to mild or from Visit 2 severity of moderate to none after treatment as measured by the Investigator's live assessment.
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: ITT Population; N'= number of subjects with an Investigator's live assessment of glabellar lines at rest of moderate or severe at Baseline and with an assessment at the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 18 | 17 | 13 | 14 | 19
percentage of subjects
  ILA: Day 8 (N'=18,17,13,14,19) | 5.6 | 5.9 | 23.1 | 21.4 | 10.5
  ILA: Day 15 (N'=18,17,13,14,18) | 5.6 | 17.6 | 23.1 | 21.4 | 16.7
  ILA: Day 29 (N'=18,17,13,14,19) | 0 | 11.8 | 23.1 | 28.6 | 21.1
  ILA: Day 57 (N'=17,16,13,14,19) | 5.9 | 18.8 | 15.4 | 21.4 | 15.8
  ILA: Day 85 (N'=18,17,12,14,19) | 0 | 17.6 | 16.7 | 7.1 | 15.8
  ILA: Day 113 (N'=18,17,13,14,19) | 0 | 5.9 | 23.1 | 14.3 | 5.3

10. Secondary Outcome: Percentage of Subjects With a Reduction of Two or More Grades in the Severity of Glabellar Lines at Maximum Frown as Measured by the Subject's Self-assessment
Description: A reduction of two or more grades in the severity of glabellar lines at maximum frown was a change from Visit 2 severity of glabellar lines from severe to mild/no wrinkles or from Visit 2 severity of moderate to no wrinkles after treatment as measured by the subjects self assessment.
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 34 | 36 | 35 | 35 | 35
percentage of subjects
  SSA: Day 8 (N'=34,36,35,35,35) | 0 | 25.0 | 42.9 | 40.0 | 34.3
  SSA: Day 15 (N'=33,36,35,35,34) | 0 | 52.8 | 57.1 | 54.3 | 47.1
  SSA: Day 29 (N'=34,36,35,33,35) | 0 | 52.8 | 60.0 | 57.6 | 57.1
  SSA: Day 57 (N'=34,35,34,34,34) | 0 | 40.0 | 52.9 | 44.1 | 47.1
  SSA: Day 85 (N'=34,35,34,32,34) | 0 | 28.6 | 29.4 | 31.3 | 29.4
  SSA: Day 113 (N'=34,36,35,34,35) | 0 | 8.3 | 22.9 | 11.8 | 17.1

11. Other Pre Specified Outcome: Number of Subjects Reporting at Least One Treatment Emergent Adverse Event During the Study
Description: Treatment Emergent Adverse Event (TEAE)
Time Frame: Up to Day 113 (±3 days)
Population: Safety Population: The safety population included all randomised subjects who received study treatment, regardless of the actual amount injected
Measure: Number; unit: participants
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 35 | 36 | 35 | 35 | 35
participants
  TEAE | 12 | 15 | 10 | 11 | 10
  Severe TEAE | 0 | 1 | 0 | 0 | 0
  Related TEAE | 5 | 6 | 4 | 4 | 2
  Related and severe TEAE | 0 | 0 | 0 | 0 | 0
  TEAE leading to withdrawal | 0 | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0 | 0
  Serious Adverse Event (SAE) | 0 | 1 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Subjects as Responders, as Measured by the Investigator's Live Assessment at Maximum Frown (Comparison With Dysport 50 U)
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: ITT Population; N'=number of subjects with assessment
Measure: Number; unit: percentage of subjects
Arm/Group | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 36 | 35 | 35 | 35
percentage of subjects
  ILA: Day 8 (N'=36,35,35,35) | 77.8 | 80.0 | 82.9 | 57.1
  ILA: Day 15 (N'=36,35,35,34) | 80.6 | 94.3 | 91.4 | 73.5
  ILA: Day 29 (N'=36,35,33,35) | 88.9 | 91.4 | 87.9 | 77.1
  ILA: Day 57 (N'=35,34,34,34) | 77.1 | 79.4 | 82.4 | 70.6
  ILA: Day 85 (N'=33,34,32,34) | 48.5 | 58.8 | 75.0 | 52.9
  ILA: Day 113 (N'=36,35,34,35) | 22.2 | 42.9 | 55.9 | 31.4

13. Secondary Outcome: Percentage of Subjects as Responders, as Measured by the Subject's Self Assessment at Maximum Frown (Comparison With Dysport 50 U)
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: ITT Population; N'=number of subjects with assessment
Measure: Number; unit: percentage of subjects
Arm/Group | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 36 | 35 | 35 | 35
percentage of subjects
  SSA: Day 8 (N'=36,35,35,35) | 66.7 | 65.7 | 74.3 | 57.1
  SSA: Day 15 (N'=36,35,35,34) | 80.6 | 82.9 | 80.0 | 73.5
  SSA: Day 29 (N'=36,35,33,35) | 91.7 | 85.7 | 81.8 | 82.9
  SSA: Day 57 (N'=35,34,34,34) | 80.0 | 67.6 | 82.4 | 73.5
  SSA: Day 85 (N'=35,34,32,34) | 57.1 | 47.1 | 62.5 | 41.2
  SSA: Day 113 (N'=36,35,34,35) | 36.1 | 34.3 | 52.9 | 28.6

14. Secondary Outcome: Percentage of Subjects as Responders, as Measured by the Investigator's Live Assessment at Rest (Comparison With Dysport 50 U)
Time Frame: Days 8, 15, 29, 57, 85 and 113
Population: ITT Population; N'=number of subjects with an Investigator's live assessment of glabellar lines at rest of moderate or severe at Baseline and with an assessment at the given post-Baseline visit
Measure: Number; unit: percentage of subjects
Arm/Group | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Number analyzed (Participants) | 17 | 13 | 14 | 19
percentage of subjects
  ILA: Day 8 (N'=17,13,14,19) | 70.6 | 76.9 | 71.4 | 63.2
  ILA: Day 15 (N'=17,13,14,18) | 70.6 | 92.3 | 78.6 | 72.2
  ILA: Day 29 (N'=17,13,14,19) | 82.4 | 76.9 | 85.7 | 84.2
  ILA: Day 57 (N'=16,13,14,19) | 81.3 | 76.9 | 78.6 | 84.2
  ILA: Day 85 (N'=17,12,14,19) | 82.4 | 75.0 | 64.3 | 68.4
  ILA: Day 113 (N'=17,13,14,19) | 52.9 | 53.8 | 57.1 | 52.6

15. Secondary Outcome: Percentage of Subjects as Responders at Day 29 by the Investigator's Live Assessment and by Subject's Self Assessment of Glabellar Lines at Maximum Frown (Assay Sensitivity)
Time Frame: Day 29
Population: ITT Population; N'=number of subjects with an assessment at Day 29
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Dysport 50 U
Number analyzed (Participants) | 34 | 35
percentage of subjects
  ILA: (N'=34,35) | 0 | 77.1
  SSA: (N'=34,35) | 2.9 | 82.9

ADVERSE EVENTS:
Time Frame: Up to Day 113 (±3 days)
Groups:
- Dysport 50 U: Botulinum type A toxin ((Azzalure), Intramuscular injections on Day 1 (total injection volume of 0.25 ml divided into five intramuscular injections of 0.05 mL per injection each of which was injected into five pre-defined sites across the glabellar region) (single treatment cycle)
Arm/Group | Placebo | Dysport NG 20 U | Dysport NG 50 U | Dysport NG 75 U | Dysport 50 U
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/36 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 12/35 | 14/36 | 10/35 | 11/35 | 10/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | Dysport NG 20 U (N=36) | Dysport NG 50 U (N=35) | Dysport NG 75 U (N=35) | Dysport 50 U (N=35)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | Dysport NG 20 U (N=36) | Dysport NG 50 U (N=35) | Dysport NG 75 U (N=35) | Dysport 50 U (N=35)
Headache (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3) | 2 (3) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site anaesthesia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laparoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No